CLINICAL TRIAL: NCT03391297
Title: Shortened Prolonged Exposure Therapy for Chronic PTSD: A Systematic Case Study
Brief Title: Shortened Prolonged Exposure Therapy for Chronic PTSD in Taiwanese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yi-Jen Su, Assistant Professor, Chang Gung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOST 106-2628-H-182-001-SS2
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; prolonged exposure; posttraumatic growth
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prolonged exposure therapy (PE), a specific exposure therapy for PTSD, has been proved an effective treatment for PTSD. PE usually consists of 10-15 individual sessions. Treatment includes psychoeducation, in vivo exposure (i.e., confronting trauma-related situations and objects that are being avoided), imaginal exposure (i.e., revisiting and recounting traumatic memory) followed by processing (discussing the experience of revisiting the trauma memory, with a focus on new learning and changed beliefs or perspectives).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60-minute Prolonged Exposure Therapy (Experimental): This condition is a modified version of Prolonged Exposure Therapy for PTSD. It consists of weekly 60-minute sessions, with at least 20 minutes imaginal exposure.
  Interventions: Behavioral: Prolonged Exposure Therapy
- 90-minute Prolonged Exposure Therapy (Active Comparator): This condition is standard Prolonged Exposure Therapy. It consists of 10 to 15 weekly sessions, each lasting about 90 minutes, with 40-60 minutes imaginal exposure.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — PE consists of 10-15 treatment sessions. Treatment includes psychoeducation, in vivo exposure (i.e., confronting trauma-related situations and objects that are being avoided), imaginal exposure (i.e., revisiting and recounting traumatic memory) followed by processing (discussing the experience of revisiting the trauma memory, with a focus on new learning and changed beliefs or perspectives).

SUMMARY:
The present study aimed to investigate the efficacy of 60-minute sessions of prolonged exposure (PE) for patients with posttraumatic stress disorder (PTSD) in Taiwan. A systematic case study will be employed to compare the efficacy of 60-minute PE session versus standard 90-minute session with eight Taiwanese PTSD patients. Participants will include the individuals aged 18 or older who meet a diagnosis of DSM-5 PTSD and to experience moderate to severe symptoms for at least 3 months. Those who have current substance dependence, psychosis, and acute suicidality (i.e., recent suicidal ideation with intent and plan) will be excluded. Participants will receive 10-15 weekly session of PE treatment with 60- or 90-minute sessions. The investigators hypothesized that: (a) 60-minute PE is as effective as 90-minute PE in reducing PTSD and depressive symptoms as well as in promoting posttraumatic growth (PTG); and (b) the treatment gains will be maintained at 3-month follow-up.

DETAILED DESCRIPTION:
Background: Posttraumatic stress disorder (PTSD) is a common psychological disorder following trauma and disaster. Due to the frequent occurrence of disasters induced by natural hazards, many Taiwanese people suffer from post-disaster mental health problems, suggesting the necessity of promoting evidence-based psychotherapies for PTSD in Taiwan. However, there has been little concern about this necessity over the past decades. To date, several evidence-based psychotherapies for PTSD have been developed, and prolonged exposure treatment (PE) has the largest number of studies supporting its efficacy and effectiveness. PE has been found effective with the widest range of trauma populations and has been studies across cultures. Given its strong evidence base, the investigators tested the efficacy and feasibility of PE for Taiwanese PTSD patients. It is noted that the original length of PE session is 90 minutes, which is difficult to get reimbursement by insurance and may prevent mental health professionals to use PE. Recent researchers shortened the length of PE session to 60 minutes and found its efficacy was non-inferior to standard 90-minute PE session (Nacasch et al., 2015; van Minnen & Foa, 2006). Accordingly, this study aims to examine the efficacy of 60-minute PE sessions versus standard 90-minute session for patients with PTSD in Taiwan.

Study Hypothesis: (a) 60-minute PE session is as effective as 90-minute PE session in reducing PTSD and depressive symptoms as well as in promoting posttraumatic growth (PTG); and (b) the treatment gains will be maintained at 3-month follow-up. A systematic case study will be employed to test the hypotheses.

Participants: Participants will include eight individuals aged 18 or older who meet a diagnosis of DSM-5 PTSD and to experience moderate to severe symptoms for at least 3 months. Those who have current substance dependence, psychosis, and acute suicidality (i.e., recent suicidal ideation with intent and plan) will be excluded.

Study Design: All enrolled participants will attend 10-15 weekly 60- or 90-minute PE sessions. Independent evaluators will assess PTSD diagnosis using the PTSD Symptoms Scale Interview for DSM-5 (PSSI-5) at pre- and post-treatment and at the three-month follow-up. Psychiatric comorbidity will be assessed using the MINI 7.0.2 at pretreatment. Participants will complete the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5), Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), Posttraumatic Cognitions Inventory (PTCI), and Posttraumatic Growth Inventory -Extended version (PTGI-X) at pre- and post-treatment and at the three-month follow-up. The PDS-5 and BDI-II will also be administered every two weeks during treatment.

Statistical Analysis: The nonparametric tests will be used given the small sample size. Wilcoxon signed-rank test will be conducted to test pre-post differences. Mann-Whitney U test will be conducted examine whether 60-minute PE session is as effective as 90-minute PE session in reducing PTSD and depressive symptoms as well as increasing PTG at post-treatment and three-month follow-up.

Expected Outcome: The investigators except that shortened PE will result in substantial improvement in PTSD and depressive symptoms in patients with PTSD in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of DSM-5 PTSD, with moderate to severe symptoms for at least 3 months

Exclusion Criteria:

* organic mental disorder, current substance dependence, psychosis, acute suicidality (i.e., suicidal ideation with intent and plan), and severe dissociation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-01-10 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Interviewer-assessed PTSD diagnosis and symptoms | Pre-treatment through three-month follow-up
  as measured by the Chinese version of the PTSD Symptoms Scale Interview for DSM-5 (PSSI-5) (Foa et al., 2016). The tota score ranged from 0 to 80, with higher scores indicating greater PTSD symptoms.

SECONDARY OUTCOMES:
Self-reported PTSD symptoms | Pre-treatment through three-month follow-up
  as measure by the Chinese version of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5; Foa et al., 2016). The tota score ranged from 0 to 80, with higher scores indicating greater PTSD symptoms.
Self-reported depressive symptoms | Pre-treatment through three-month follow-up
  as measure by the Chinese version of the Beck Depression Inventory-II (Beck, Steer, & Brown, 1996). The tota score ranged from 0 to 63, with higher scores indicating greater depressive symptoms.
Self-reported posttraumatic growth | Pre-treatment through three-month follow-up
  as measured by the Chinese version of the Expanded Posttraumatic Growth Inventory. The total score ranged from 0 to 75, with higher scores indicating greater trauma-related growth.
Self-reported posttraumtic negative cognitions | Pre-treatment through three-month follow-up
  as measured by the Chinese version of the Posttraumatic Cognition Inventory. The total score ranged from 33 to 231, with higher scores indicating greater posttraumatic negative cognitions.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Su, Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Graduate Institute of Behavioral Sciences, Chang Gung University, Taoyuan District, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No